CLINICAL TRIAL: NCT05738434
Title: A Randomized, Controlled, Multicenter Clinical Study of Camrelizumab in Combination With Apatinib Mesylate and Chemotherapy Versus Camrelizumab Plus Chemotherapy in the First-line Treatment of Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Camrelizumab in Combination With Apatinib Mesylate Plus Short-course Chemotherapy for Advanced ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-EC-II-014
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Cancer by AJCC V8 Stage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-course Chemotherapy (Experimental)
  Interventions: Drug: Camrelizumab+Apatinib+Chemotherapy→Camrelizumab+Apatinib
- Chemotherapy (Active Comparator)
  Interventions: Drug: Camrelizumab+Chemotherapy→Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab+Apatinib+Chemotherapy→Camrelizumab+Apatinib — camrelizumab 200 mg, i.v. d1,q3w; apatinib 250 mg, p.o. qd,q3w; cisplatin 25 mg/m2, i.v. d1-d3,q3w; According to investigator' choice： paclitaxel 135~150 mg/m2, i.v. d1,q3w; paclitaxel-albumin 150~180 mg/m2, i.v. d1,q3w. up to 4 cycles and sequential maintenance therapy： camrelizumab 200 mg, i.v. d1,q3w; apatinib 250 mg, p.o. qd,q3w
  Arms: Short-course Chemotherapy
Drug: Camrelizumab+Chemotherapy→Camrelizumab — camrelizumab 200 mg, i.v. d1,q3w; cisplatin 25 mg/m2, i.v. d1-d3,q3w; According to investgator' choice： paclitaxel 175 mg/m2, i.v. d1,q3w; paclitaxel-albumin 200 mg/m2, i.v. d1,q3w up to 6 cycles and sequential maintenance therapy： camrelizumab 200 mg, i.v. d1,q3w;
  Arms: Chemotherapy

SUMMARY:
To evaluate the efficacy and safety of patients with advanced esophageal squamous cell carcinoma treated with camrelizumab combined with Apatinib mesylate plus short-course chemotherapy versus standard chemotherapy in first line

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75, male or female;
* 2. Esophageal squamous cell carcinoma that is histologically or cytologically confirmed as unresectable locally advanced/recurrent (unable to receive radical treatment such as radical chemoradiotherapy or radical radiotherapy) or distant metastasis;
* 3. No previous systematic antitumor therapy. For patients who received neoadjuvant/adjuvant and radical concurrent chemoradiotherapy, the time from the last chemotherapy to recurrence or progression more than 6 months can be screened;
* 4. According to the efficacy evaluation criteria for solid tumors (RECIST 1.1), there should be at least one measurable lesion (esophageal and other cavity structures cannot be used as measurable lesions), and the measurable lesions should not have received local treatment such as radiotherapy (lesions located within the previous radiotherapy area can also be selected as target lesions if it is confirmed to progress);
* 5. Agree to provide tissue samples for biomarker (such as PD-L1) analysis. Recently obtained tissues are preferred. Patients who cannot provide recently obtained tissues can provide 5-8 paraffin sections of 3-5 μm thickness for archival storage;
* 6. ECOG PS: 0 ~ 1;
* 7. Swallowing pills normally;
* 8. Expected survival ≥12 weeks;
* 9. The functions of vital organs meet the following requirements (no drugs with blood components and cell growth factors are allowed to be used within 14 days before the first use of the study drug);

  1. Absolute count of neutrophils (ANC) ≥1.5×109/L
  2. Platelet ≥90×109/L;
  3. Hemoglobin ≥90g/L;
  4. Serum albumin ≥28g/L;
  5. Total bilirubin ≤1.5 × ULN, ALT, AST, and/or AKP≤2.5 × ULN; If liver metastasis is present, ALT and/or AST≤5 × ULN; If there is liver metastasis or bone metastasis AKP≤5 × ULN;
  6. Serum creatinine ≤1.5 × ULN or creatinine clearance > 60 mL/min (Cockcroft-Gault);
  7. Activated partial thromboplastin time (APTT) and International Normalized ratio (INR) ≤1.5 × ULN (for stable dose anticoagulant therapy such as low molecular weight heparin or warfarin and INR within the expected treatment range of anticoagulants can be screened)
* 10. Fertile female subjects and male subjects whose partners are women of childbearing age, A medically approved contraceptive (such as an intrauterine device, contraceptive or condom) is required during the study treatment period and at least 2 months after the last use of carrilizumab/Apatinib mesylate and at least 6 months after the last use of chemotherapy;
* 11. The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* 1. BMI < 18.5 kg/m2 or weight loss ≥10% within 2 months prior to screening (while the effect of large amounts of abdominal and thoracic fluids on body weight should be considered);
* 2. Active hemoptysis occurred within 3 weeks before the first administration of the study drug, or tumor hemorrhage occurred within 2 weeks before the first administration of the study intervention;
* 3. Patients with tumors assessed by the investigator to have invaded adjacent organs of the esophageal lesion (such as the aorta or respiratory tract) and had a high risk of bleeding or fistula during the study;
* 4. Previous history of gastrointestinal perforation and/or fistula or recent (within 3 months before randomization) history of intestinal obstruction or imaging and clinical symptoms suggestive of intestinal obstruction;
* 5. Subjects who have had esophageal stents implanted or are evaluated for needing esophageal stents implanted;
* 6. Patients with clinical symptoms of pleural effusion, pericardial effusion or ascites who need puncture or drainage or who have received drainage for treatment within 1 month before randomization;
* 7. Have high blood pressure that is not well controlled by antihypertensive medications (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
* 8. A history of allergies to monoclonal antibodies, any component of Camrelizumab, Apatinib mesylate and its excipients, paclitaxel, albumin paclitaxel and cisplatin;
* 9. Received any of the following medical treatment:

  1. Received any investigational drug within 4 weeks prior to initial use of the investigational drug;
  2. Enrolling in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up;
  3. Receiving the last dose of anticancer therapy (including radiotherapy, etc.) within 4 weeks or less before the first use of the study drug;
  4. Subjects who required systemic treatment with corticosteroids (> 10 mg daily equivalent of prednisone) or other immunosuppressant within 2 weeks prior to initial use of the study drug, except for corticosteroids for local esophageal inflammation and prevention of allergy, nausea, and vomiting. In the absence of active autoimmune disease, inhaled or topical steroid and adrenocortical hormone replacement at doses > 10mg/ day of prednisone efficacy dose are permitted;
  5. Those who have received anti-tumor vaccine or have received live vaccine within 4 weeks prior to the first administration of the study drug;
  6. Major surgery or severe trauma within 4 weeks prior to initial use of the study drug;
* 10. The toxicity of previous antitumor therapy has not recovered to ≤CTCAE Grade 1 (except hair loss) or the level specified by inclusion/exclusion criteria;
* 11. Patients with central nervous system metastasis;
* 12. History of active autoimmune diseases, autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitaries, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Except for patients with vitiligo or asthma/allergies from childhood that have recovered and require no intervention as adults; Autoimmune mediated hypothyroidism treated with a steady dose of thyroid replacement hormone; Type 1 diabetes using a steady dose of insulin;
* 13. A history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
* 14. Subjects have poorly controlled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA Grade II or higher heart failure, (2) unstable angina pectoris, (3) previous myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias that are not well controlled without clinical intervention or after clinical intervention;
* 15. Severe infections (CTCAE > Grade 2), such as severe pneumonia, bacteremia, and infection complications requiring hospitalization, occurred within 4 weeks prior to the first use of the study drug; Baseline chest imaging indicated active pulmonary inflammation, signs and symptoms of infection within 2 weeks prior to initial use of the study drug, or the need for oral or intravenous antibiotic treatment, except for the use of prophylactic antibiotics;
* 16. History of interstitial lung disease (except radiation pneumonia without hormone therapy) and non-infectious pneumonia;
* 17. Patients with active tuberculosis infection identified by medical history or CT examination, or with a history of active tuberculosis infection within 1 year prior to enrollment, or with a history of active tuberculosis infection more than 1 year ago but without formal treatment;
* 18. Subjects had active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (HCV antibody positive and HCV-RNA above the assay limit);
* 19. Bleeding symptoms of significant clinical significance or definite bleeding tendency, such as digestive tract bleeding, hemorrhagic ulcer or vasculitis, have occurred within 3 months before randomization. If stool occult blood is positive in baseline period, review can be conducted; if it is still positive after review, combined with clinical judgment, gastroscopy should be performed if necessary;
* 20. Arteriovenous thrombosis events occurring within 6 months prior to randomization, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, and cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. Superficial vein thrombosis could be included after being determined by the researchers;
* 21. Known hereditary or acquired bleeding and thrombotic tendencies (e.g. haemophiliacs, coagulation disorders, thrombocytopenia, etc.);
* 22. With active ulcers, unhealed wounds or with fractures;
* 23. Urine routine indicated urinary protein ≥ ++ and confirmed 24-hour urinary protein volume > 1.0g;
* 24. Subjects were still using a strong CYP3A4 inducer within 2 weeks before randomization, or were still using a strong CYP3A4 inhibitor within 1 week before randomization;
* 25. Any other malignancies diagnosed within five years prior to the first use of the study drug, other than those with a low risk of metastasis and death (5-year survival > 90%), such as basal or squamous cell skin cancer or carcinoma in situ of the cervix after adequate treatment;
* 26. Pregnant or lactating women;
* 27. In the investigator's judgment, the subjects had other factors that might have led to their being forced to terminate the study, such as other serious medical conditions (including mental illness) requiring concomitant treatment, serious abnormalities in laboratory test values, or family or social factors that might have affected the subjects' safety or the circumstances in which the study data were collected.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS[Progression-Free Survival] | up to 2 year
  Time from randomization to first radiographic disease progression (RECIST 1.1 criteria) or death, whichever occurs first.

SECONDARY OUTCOMES:
OS[Overall Survival] | up to 2 year
  Time from randomization to the subject's death. At the end of the study, if the subject is still alive, the last known date of survival of the subject will be the date of deletion.
ORR[Objective Response Rate] | up to 1 year
  Proportion of subjects in the analysis population who achieved complete response (CR) or partial response (PR) based on RECIST 1.1 criteria.
DCR[Disease Control Rate] | up to 1 year
  Proportion of subjects in the analysis population who achieved complete response (CR) , partial response (PR) or stable disease(SD) based on RECIST 1.1 criteria.
TTR[Time to response] | up to 1 year
  Time from randomization to firstly achieve CR or PR based on RECIST 1.1 criteria.
DoR[Duration of response] | up to 2 year
  For subjects who achieved remission, the time from first achieving CR or PR to disease progression or death, whichever occurred earlier.
AEs[Adverse events] | up to 2 year
  The incidence and severity of adverse events (AE) and serious adverse events (SAE) were determined according to NCI-CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, phD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No